CLINICAL TRIAL: NCT02419599
Title: The Effect of Standard Versus High Energy Density, Low Volume Oral Nutritional Supplements in Children Requiring Nutritional Support - a Pilot Trial
Brief Title: High vs Standard Energy Children's Drink Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FC125
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Growth Failure
MeSH Terms: conditions — Failure to Thrive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): The group who will receive high energy density, low volume oral nutritional supplement, to be taken for 4 weeks (28 days)
  Interventions: Other: HE ONS
- Group B (Active Comparator): The group who will receive the standard energy density oral nutritional supplement, to be taken for 4 weeks (28 days)
  Interventions: Other: SE ONS

INTERVENTIONS:
Other: HE ONS — High energy density, low volume oral nutritional supplement (HE ONS) in addition to appropriate nutritional management
  Arms: Group A
Other: SE ONS — Standard energy density oral nutritional supplement (SE ONS) in addition to appropriate nutritional management
  Arms: Group B

SUMMARY:
This study is a pilot trial investigating the effects of a high energy drink for children, in comparison to standard energy drink for children.

DETAILED DESCRIPTION:
A four week, multi-centre, randomised controlled trial investigating the effects of a high energy density, low volume oral nutritional supplement versus standard energy density oral nutritional supplements in children aged 1-12yrs old requiring nutritional support. Fifty eligible children will be recruited and randomised to receive either the high energy density oral nutritional supplement or the standard energy density oral nutritional supplement for four weeks. The primary outcome is nutrient intake, with secondary outcomes of compliance, tolerance, acceptability, anthropometry and safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 1-12yrs
* Faltering growth and/or requiring oral nutritional supplements to meet nutritional requirements
* Expected to receive at least one bottle of the study product per day
* Able to take study products orally during the study period
* Written informed consent from parent/carer

Exclusion Criteria:

* Requirement for 100% of their nutrition via enteral tube and/or parenteral feeding.
* Children with major hepatic or renal dysfunction
* Children with galactosaemia or severe lactose intolerance
* Requirement for elemental or semi-elemental feeds
* Investigator concern around willingness/ability of child/parent/carer to comply with protocol requirements
* Participation in other studies within 2 weeks of study

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Nutrient intake | 4 weeks (28 days)
  Dietary intake, including the intake of all foods and fluids, will be recorded and analysed throughout the study.

SECONDARY OUTCOMES:
Compliance: Compliance with oral nutritional supplements in Group A and Group B; how much of the oral nutritional supplement is taken in comparison to the amount advised by the Dietitian. | 4 weeks (28 days)
Tolerance: How well the child tolerates the oral nutritional supplements (including changes to gastrointestinal symptoms) | 4 weeks (28 days)
Acceptability: How acceptable the oral nutritional supplement is to the child and their parent/carer, including taste, texture, ease of use, etc. | 4 weeks (28 days)
Anthropometry | 4 weeks (28 days)
  Changes to weight, height and head circumference in children less than 2yrs of age.
Safety assessed by adverse events, to be recorded throughout study. | 4 weeks (28 days)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hubbard GP, Fry C, Sorensen K, Casewell C, Collins L, Cunjamalay A, Simpson M, Wall A, Van Wyk E, Ward M, Hallowes S, Duggan H, Robison J, Gane H, Pope L, Clark J, Stratton RJ. Energy-dense, low-volume paediatric oral nutritional supplements improve total nutrient intake and increase growth in paediatric patients requiring nutritional support: results of a randomised controlled pilot trial. Eur J Pediatr. 2020 Sep;179(9):1421-1430. doi: 10.1007/s00431-020-03620-9. Epub 2020 Mar 13. PMID 32170451